CLINICAL TRIAL: NCT04674111
Title: Vortex - First in Human Study to Evaluate the Feasibility, Safety, Clinical and Technical Success of the Vortex Temporary Percutaneous, Transvalvular Circulatory Support System (Vortex System)
Brief Title: Vortex - Temporary Percutaneous, Transvalvular Circulatory Support System Feasibility Study
Acronym: Vortex-FIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S2465
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: Mechanical circulatory support; High risk percutaneous coronary intervention (HR PCI)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, single-arm feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vortex Feasibility Study (Vortex FIH) (Experimental): Vortex - First in Human Study to Evaluate the Feasibility, Safety, Clinical and Technical Success of the Vortex Temporary Percutaneous, Transvalvular Circulatory Support System (Vortex System)
  Interventions: Device: Temporary Percutaneous Transvalvular Circulatory Support System (Vortex System)

INTERVENTIONS:
Device: Temporary Percutaneous Transvalvular Circulatory Support System (Vortex System) — The Vortex System is intended to provide temporary circulatory support in subjects undergoing elective high-risk percutaneous coronary intervention (HR-PCI).

SUMMARY:
Vortex - First in Human study to evaluate the feasibility, safety, clinical and technical success of the Vortex temporary percutaneous, transvalvular circulatory support system (Vortex System)

ELIGIBILITY:
Inclusion Criteria:

A subject will be considered for enrolment in the study if all of the following inclusion criteria are met, provided no exclusion criteria are met:

IC1. Subject provides signed informed consent. IC2. Subject is ≥ 18 years and < 90 years of age.

IC3 Subject is indicated for NON-emergent PCI of at least one de novo or restenotic lesion in a native coronary vessel or coronary artery bypass graft (CABG) and has left ventricular ejection fraction (LVEF) ≤ 50% with the following:

* Unprotected left main -OR-
* Last remaining vessel -OR-
* Three vessel disease (≥ 50% diameter stenoses by visual estimate or total occlusion)

Exclusion Criteria:

A subject will be excluded from the study if any of the following exclusion criteria are met:

EC1. Subject has had ST-elevation myocardial infarction (STEMI) within 24 hours.

EC2. Subject has had pre-procedure cardiac arrest requiring cardiopulmonary resuscitation (CPR) within 24 hours of enrollment.

EC3. Subject is in shock, defined as follows:

* Cardiac index (CI) < 2.2 L/min/m2 and pulmonary capillary wedge pressure (PCWP) > 15 mmHg -AND-
* Hypotension (systolic blood pressure < 90 mmHg for > 30 minutes) -OR-
* Need for supportive measures (i.e., inotropes or mechanical support) to maintain systolic blood pressure ≥ 90 mmHg and end organ hypoperfusion (cool extremities or urine < 30 mL/hour and a heart rate > 60 beats per minute) EC4. Subject has left ventricular mural thrombus. EC5. Subject has a prosthetic aortic valve. EC6. Subject has pericarditis or constrictive heart disease (constrictive pericarditis or restrictive cardiomyopathy).

EC7. Subject has moderate or greater aortic valve stenosis or moderate or greater aortic valve insufficiency (by echocardiographic assessment, graded as ≥ 2+).

EC8. Subject has abnormalities of the aorta that preclude safe delivery of the device, including severe calcification, tortuosity, aneurysm, or prior surgery.

EC9. Subject has peripheral vessel disease (PVD) preventing passage of the device (e.g., calcification, small caliber) or tortuosity that would preclude safe placement of the 16 Fr introducer sheath.

Note: Minimum required vessel diameter is > 5.5 mm. EC10. Subject has advanced renal dysfunction (AKIN Stage 3). EC11. Subject has a history of liver dysfunction (Childs Class C) with elevation of liver enzymes and bilirubin > 3× upper limit of normal (ULN) or international normalization ratio (INR) ≥ 2.

EC12. Subject has had a recent (within 1 month) stroke or TIA. EC13. Subject has known hypersensitivity to intravenous contrast agents that cannot be adequately pre-medicated or has known hypersensitivity to heparin, aspirin, ADP receptor inhibitors or nitinol.

EC14. Subject has current or a history of heparin induced thrombocytopenia (HIT).

EC15. Subject has uncorrected abnormal coagulation or platelet count ≤ 75,000/mm³ or INR ≥ 2.0.

EC16. Subject has significant right heart failure (right atrial pressure [RAP] > 15 mmHg, right ventricular stroke work index [RVSWI] < 0.30 mmHg·L/m², pulmonary vascular resistance [PVR] > 3.6 Woods units).

EC17. Subject requires mechanical ventilation. EC18. Subject has an atrial or ventricular septal defect (including post-infarct ventricular septal defect [VSD]).

EC19. Subject has left ventricular rupture. EC20. Subject has cardiac tamponade. EC21. Subject has severe pulmonary disease (FEV1 < 1L). EC22. Subject has sustained or non-sustained ventricular tachycardia. EC23. Subject is breast feeding or is pregnant.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Antony Walton, MBBS, Principal Investigator — The Alfred
Locations (2):
- The Alfred Hospital, Melbourne, Victoria, Australia
- Skane University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Vortex Feasibility Study (Vortex FIH): Vortex - First in Human Study to Evaluate the Feasibility, Safety, Clinical and Technical Success of the Vortex Temporary Percutaneous, Transvalvular Circulatory Support System (Vortex System)
  Temporary Percutaneous Transvalvular Circulatory Support System (Vortex System): The Vortex System is indicated to provide temporary circulatory support in subjects undergoing elective high-risk percutaneous coronary intervention (HR-PCI).
Period: Overall Study
Arm/Group | Vortex Feasibility Study (Vortex FIH)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vortex Feasibility Study (Vortex FIH)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.6 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Technical Success
Description: Successful delivery of the device to the correct anatomical position and successful operation and removal of the Vortex circulatory support system during high-risk PCI procedure.
Time Frame: Technical success is measured during the procedure. Procedure time varies by patient and is measured from 1st vascular puncture for sheath insertion to vascular closure post sheath removal. Mean procedure time was 116.0 minutes (70.0 min, 148.0 max).
Measure: Count of Participants; unit: Participants
Arm/Group | Vortex Feasibility Study (Vortex FIH)
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: Number of Participants With Clinical Success
Description: No conversion to open heart surgery during the high-risk PCI procedure and no in-hospital mortality.
Time Frame: Clinical success is measured during the procedure. Procedure time varies by patient and is measured from 1st vascular puncture for sheath insertion to vascular closure post sheath removal. Mean procedure time was 116.0 minutes (70.0 min, 148.0 max).
Measure: Count of Participants; unit: Participants
Arm/Group | Vortex Feasibility Study (Vortex FIH)
Number analyzed (Participants) | 5
Participants | 5

ADVERSE EVENTS:
Time Frame: Through 72 hours post index procedure or at hospital discharge (whichever comes first)
Arm/Group | Vortex Feasibility Study (Vortex FIH)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortex Feasibility Study (Vortex FIH) (N=5)
Hypotension (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vortex Feasibility Study (Vortex FIH) (N=5)
Decrease in Hemoglobin (Blood and lymphatic system disorders) | 2 (2)
Arterial hemorrhage (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-05-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT04674111/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT04674111/SAP_001.pdf